CLINICAL TRIAL: NCT07282067
Title: A Retrospective Study to Assess the Efficacy of PEMF Treatment in Ankle Fusion
Brief Title: Orthofix PhysioStim PEMF Ankle Fusion Retrospective
Acronym: PSAF
Status: Active, not recruiting | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-PSAF-24
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Ankle Fusion; Hindfoot Arthrodesis; Ankle Arthrodesis; Tibiotalar Arthrodesis
Keywords: ankle; tibiotalar; PEMF; hindfoot; pulsed electromagnetic fields; Orthofix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- PEMF use adjunct to ankle/hindfoot fusion: This group will include subjects where PhysioStim (PEMF) is used adjunctively to an ankle/hindfoot fusion procedure.
  Interventions: Device: Pulsed electromagnetic field (PEMF) stimulation
- PEMF use for failed ankle/hindfoot fusion: This group will include subjects where PhysioStim (PEMF) is used to treat a failed ankle/hindfoot fusion procedure.
  Interventions: Device: Pulsed electromagnetic field (PEMF) stimulation
- Ankle/hindfoot fusion, no device (Control): This group will include subjects where PhysioStim (PEMF) is NOT used adjunctively to an ankle/hindfoot fusion procedure. Subjects will be identified as those indicated to receive PEMF, but did not due to reasons such as insurance denial, patient declined to use the device, etc.
  Interventions: Other: Control
- Failed ankle/hindfoot fusion, no device (Control): This group will include subjects where PhysioStim (PEMF) is NOT used to treat a failed ankle/hindfoot fusion procedure. Subjects will be identified as those indicated to receive PEMF, but did not due to reasons such as insurance denial, patient declined to use the device, etc.
  Interventions: Other: Control

INTERVENTIONS:
Device: Pulsed electromagnetic field (PEMF) stimulation — Subjects treated with PEMF with be directed to use the device for 3 hours per day, up to 6 months or until no longer needed.
  Groups: PEMF use adjunct to ankle/hindfoot fusion; PEMF use for failed ankle/hindfoot fusion
Other: Control — Control (no PEMF)
  Groups: Ankle/hindfoot fusion, no device (Control); Failed ankle/hindfoot fusion, no device (Control)

SUMMARY:
This study examines the effect of using the PhysioStim bone growth stimulator on subjects undergoing treatment for ankle and hindfoot fusion surgery.

DETAILED DESCRIPTION:
The objective of this investigation is to study the effect of using adjunctive PEMF treatment (via PhysioStim) in subjects undergoing ankle fusion, and also as nonoperative treatment for failed ankle fusion. The sponsor hypothesizes that use of PhysioStim will result in higher rates of fusion compared to that of control. In addition to analyzing the primary endpoint, the study will collect safety information to confirm the favorable safety profile established in prior device usage.

ELIGIBILITY:
Inclusion Criteria:

* Condition requiring ankle fusion surgery or nonoperative treatment for failed ankle fusion
* Age 23 years or older
* Subjects must have a minimum of 6 months follow-up data or evidence of fusion, whichever occurs first

Exclusion Criteria:

* Subject is a prisoner

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will be males and females who underwent an ankle fusion procedure and were at least 23 years of age at the time of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Radiographic fusion rate at 6 months post treatment | 6 months from the start of treatment
  Fusion rate (# subjects fused / # total evaluable subjects) based on radiographic assessment.

OTHER OUTCOMES:
Secondary surgeries | For the period 12 months following the start of treatment
  Rate of secondary surgeries (# subjects requiring additional surgeries / # eligible subjects)
Safety endpoints | For the period 12 months following the start of treatment
  Incidence of device and procedure-related Adverse Events (AEs) and Serious Adverse Events (SAEs) through 12 months post-treatment.
Pain (NPRS) (0-100) | Multiple, up to 12 months
  Pain reduction using Numerical Pain Rating Scale (NPRS) will be reported at multiple time points, as available. 0-100 pain scale is used where 100 is maximum pain.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Arizona Foot Health, Phoenix, Arizona
  - Phoenix Foot and Ankle Institute, Scottsdale, Arizona
  - OrthoArizona, Scottsdale, Arizona
  - Byron COllier DPM, Inc, Pismo Beach, California
  - East Village Foot and Ankle, Des Moines, Iowa
  - Precision Orthopedics and Sports Medicine, Laurel, Maryland
  - OrthoCarolina Research Institute, Inc, Charlotte, North Carolina
  - Lone Star Orthopaedic and Spine Specialists, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Undecided